CLINICAL TRIAL: NCT05281094
Title: A Phase 2b, Double-blind, Randomized, Multi-site, Placebo-controlled Trial to Evaluate the Efficacy, Safety and Immunogenicity of Intramuscular HIL-214 Norovirus Vaccine in Healthy Children 5 Months of Age at Initial Vaccination
Brief Title: Efficacy and Safety of Two Doses of HIL-214 in Children
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: HilleVax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-212
Record Dates: First submitted 2022-02-17; First posted 2022-03-16 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): One dose of placebo on Day 1 and one dose of placebo between Day 28 and Day 56.
  Interventions: Biological: Placebo
- Experimental (Experimental): One dose of HIL-214 on Day 1 and one dose of HIL-214 between Day 28 and Day 56.
  Interventions: Biological: HIL-214

INTERVENTIONS:
Biological: HIL-214 — 2 injections - given on Day 1 and the second given between Day 29 - Day 57
  Arms: Experimental
Biological: Placebo — 2 injections - given on Day 1 and the second given between Day 29 - Day 57
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled study that is being done to evaluate the safety and effectiveness of two doses of the HIL-214 vaccine compared to a placebo. The study will enroll 3000 children who will be 5 months of age at the time of the first dose study vaccine. The second dose of study vaccine will be given 28 days after the first dose.

DETAILED DESCRIPTION:
Noroviruses have emerged as the single most significant cause of gastroenteritis in both middle-high income countries and low resource settings worldwide. Those most at risk of severe illness include the very young, the elderly and immunocompromised individuals. Noroviruses are highly infectious, highly resistant to environmental conditions, and have multiple routes of transmission including person-to-person, food-borne and contaminated surfaces. Noroviruses can cause acute, mild to severe illness characterized by vomiting, diarrhea, fever, dehydration and abdominal pain, representing a significant burden to public health. The clinical presentation in adults and older children is similar. While mortality due to acute gastroenteritis (AGE) caused by norovirus in the pediatric population is rare in industrialized countries, it is more common in developing countries. Although potentially a cause for hospitalization in very young children, there are fewer cases during the first 6 months of life possibly due to the protection offered by maternal antibodies from trans-placental transfer and in breast milk. In addition, norovirus infections have significant socioeconomic impact on hospitals, schools, day care centers and other closed settings. As the burden of rotavirus in children decreases due to successful rotavirus vaccination programs in infants, norovirus infections are increasingly recognized as the primary cause of AGE in many countries around the world.

ELIGIBILITY:
Inclusion Criteria

* The subject should be 5 months of age (within plus or minus 14 days) male or female
* Children who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator
* The subject's LAR signs and dates a written, informed consent form (ICF) and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements
* Children whose LARs can and are willing to comply with trial procedures and are available for the duration of follow-up

Exclusion Criteria

* Clinically significant abnormality in growth by height, weight, or head circumference (according to local guidelines)
* Gastrointestinal abnormalities or any chronic gastrointestinal disease, including any uncorrected congenital malformation of the gastrointestinal tract according to medical history and/or physical examination
* Known hypersensitivity or allergy to any of the investigational vaccine components (including excipients)
* Any clinically significant active infection (as assessed by the investigator) or temperature ≥38.0°C (>100.4°F), within 3 days of intended trial vaccination
* Any serious chronic or progressive disease according to the judgment of the investigator (e.g., cardiac, renal or hepatic disease)
* Individuals with history of, e.g., convulsions/febrile convulsions, or any illness, that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the subjects due to participation in the trial
* Known or suspected impairment/alteration of immune function
* Subjects with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time
* Subjects who received or are scheduled to receive any other vaccines within 14 days (for inactivated vaccines and oral polio vaccine) or 28 days (for other live vaccines) before or after any dose of trial vaccine
* Subjects participating in any clinical trial with another investigational product 30 days prior to first trial visit or intend to participate in another clinical trial at any time during the conduct of this trial
* Subjects known to be positive for or in evaluation for possible human immunodeficiency virus infection
* Subject's LAR or subject's first-degree relatives involved in the trial conduct

Ages: 5 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3084 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- DM Clinical Research, Houston, Texas, United States
- Colombia (2):
  - Policlinico Social del Norte, Bogotá, Bogota D.C.
  - Cntro de Estudios en Infectologia Pediatrica (CEIP), Cali, Valle del Cauca Department
- Dominican Republic (5):
  - Hospital Pediátrico Dr. Hugo Mendoza, Santo Domingo, Nacional
  - Hospital General Regional Marcelino Velez Santana, Santo Domingo
  - CAIMED - Dominican Center for Clinical Studies, Santo Domingo
  - Clínica Cruz Jiminian, Santo Domingo
  - Fundacion Dominicana de Perinatologia Pro Bebe, Santo Domingo
- Honduras (3):
  - Demedica, San Pedro Sula
  - INVERIME - Inversiones en Investigación Medica, Tegucigalpa
  - Investigación Sin Limite, Tegucigalpa
- Panama (4):
  - CEVAXIN David, David, Chiriquí Province
  - CEVAXIN La Chorrera, La Chorrera
  - CEVAXIN 24 Decembre, Panama City
  - CEVAXIN Av. México, Panama City
- Instituto de Investigacion Nutricional, Lima, Peru
- Clinical Research Puerto Rico, Guayama, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the primary observation period of the trial (up to Visit 4) at 17 investigative sites in Panama, the Dominican Republic, Honduras, Peru, Columbia, Puerto Rico, and the United States from 28 April 2022 to 28 Dec 2023.
Pre-assignment Details: Participants were enrolled in 1 of 2 treatment arms and received 2 doses of either HIL-214, a norovirus vaccine comprising 50 µg GI.1 virus-like particle (VLP) and 150 µg GII.4c VLP, adjuvanted with 500 µg of aluminum hydroxide, or placebo.
Period: Overall Study
Arm/Group | Placebo | Experimental
Started | 1542 (6 month primary observation period, up to Visit 4) | 1542 (6 month primary observation period, up to Visit 4)
Received Two Vaccinations | 1399 | 1425
Completed | 1381 (6 month primary observation period, up to Visit 4) | 1410 (6 month primary observation period, up to Visit 4)
Not Completed | 161 | 132
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 29 | 22
Not completed — Withdrawal by Legally Authorized Representative | 122 | 103
Not completed — Death | 1 | 2
Not completed — Not pre-specified reason | 8 | 5

BASELINE CHARACTERISTICS:
Population: Modified Full-Analysis Set (mFAS): The mFAS included all participants who were randomized and received 2 doses of HIL-214 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Experimental | Total
Number analyzed (Participants) | 1399 | 1425 | 2824
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.94 (0.295) | 4.95 (0.291) | 4.95 (0.293)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 723 | 725 | 1448
  Male | 676 | 700 | 1376
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1383 | 1407 | 2790
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 1 | 0 | 1
  Race: Asian | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 14 | 9 | 23
  Race: White | 3 | 1 | 4
  Race: Other | 1302 | 1327 | 2629
  Race: More than one race | 11 | 9 | 20
  Race: Not Reported | 53 | 64 | 117
  Race: Unknown | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  Colombia | 44 | 42 | 86
  Puerto Rico | 1 | 1 | 2
  United States | 1 | 1 | 2
  Panama | 764 | 769 | 1533
  Dominican Republic | 273 | 284 | 557
  Honduras | 221 | 233 | 454
  Peru | 95 | 95 | 190
Weight [Mean (Standard Deviation); unit: kg] — Population: Weight not reported for all participants.
  kg
    number analyzed (Participants) | 1397 | 1422 | 2819
    (all) | 7.423 (0.9861) | 7.395 (0.9979) | 7.409 (0.9920)
Length [Mean (Standard Deviation); unit: cm] — Population: Length not reported for all participants.
  cm
    number analyzed (Participants) | 1397 | 1422 | 2819
    (all) | 64.16 (2.657) | 64.05 (2.731) | 64.10 (2.694)
Head circumference [Mean (Standard Deviation); unit: cm] — Population: Head circumference not reported for all participants.
  cm
    number analyzed (Participants) | 1395 | 1419 | 2814
    (all) | 42.08 (1.316) | 42.06 (1.292) | 42.07 (1.304)

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate the Efficacy of HIL-214 Vaccine Against Moderate/Severe Acute Gastroenteritis (AGE) Associated Only With GI.1 or GII.4 Norovirus Genotypes.
Description: Time to first occurrence during the primary observation period, of moderate/severe AGE case associated only with GI.1 or GII.4 norovirus genotypes. Vaccine efficacy (VE) is defined as 100% [1- (λV/λC)], where λV and λC denote the hazard rates of the primary endpoint AGE case for the HIL 214 and placebo arms, respectively. The primary endpoint AGE case is defined as at least 3 loose or liquid stools OR at least 2 or more episodes of vomiting OR 1 or more loose or liquid stools plus 1 or more vomiting episodes in any 24-hour period. The presence of norovirus in onset stool samples was assessed by RT-PCR and norovirus-positive samples were genotyped by sequencing. Samples that were positive for GI.1 or GII.4 genotypes were further analyzed for the presence of co-pathogens. VE estimates and 95% confidence intervals (CIs) are also reported.
Time Frame: The duration of the primary observation period was 6 months starting at 28 days post dose 2.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: months
Groups:
- Placebo: One dose of placebo on Day 1 and one dose of placebo between Day 29 and Day 57.
  Placebo: 2 injections - given on Day 1 and the second given between Day 29 - Day 57
- Experimental: One dose of HIL-214 on Day 1 and one dose of HIL-214 between Day 29 and Day 57.
  HIL-214: 2 injections - given on Day 1 and the second given between Day 29 - Day 57
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1399 | 1425
months | 3.07 (2.059) | 3.29 (1.746)
Statistical Analysis 1: Comparison: Placebo vs Experimental; VE is defined 100% [1- (λV/λC)], where λV and λC denote the hazard rates for the HIL-214 and placebo arms respectively, obtained via a stratified Cox proportional hazards model, using Efron's method for handling ties. The model includes a term for vaccine group and was stratified by country, whereby the United States, Dominican Republic, and Puerto Rico were considered one country. The 95% confidence interval as calculated by subtracting the confidence limits of hazard ratio from 1; Test type: Superiority; Vaccine Efficacy = 12.98, 95% CI 2-sided [-52.51 to 50.35] — . Vaccine efficacy is demonstrated if the lower limit of the 95.0% CI is above 0%

2. Secondary Outcome: To Evaluate the Efficacy of HIL-214 Vaccine Against Moderate/Severe Acute Gastroenteritis (AGE) Associated Only With Any Norovirus (GI or GII) Genogroup.
Description: Time to first occurrence during the primary observation period, of moderate/severe AGE case associated with any (GI or GII) genogroup Vaccine efficacy (VE) is defined as 100% [1- (λV/λC)], where λV and λC denote the hazard rates of the primary endpoint AGE case for the HIL 214 and placebo arms, respectively. The endpoint AGE case is defined as at least 3 loose or liquid stools OR at least 2 or more episodes of vomiting OR 1 or more loose or liquid stools plus 1 or more vomiting episodes in any 24-hour period. The presence of norovirus in onset stool samples was assessed by RT-PCR and norovirus positive samples were genogrouped by sequencing. Samples that were positive for GI or GII genogroups were further analyzed for the presence of co-pathogens. Vaccine efficacy (VE) estimates and 95% confidence intervals (CIs) are also reported.
Time Frame: The duration of the primary observation period was 6 months starting at 28 days post dose 2.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1399 | 1425
months | 3.16 (1.886) | 3.32 (1.519)
Statistical Analysis 1: Comparison: Placebo vs Experimental; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Vaccine Efficacy = 17.02, 95% CI 2-sided [-24.52 to 44.70] — Vaccine efficacy is demonstrated if the lower limit of the 95.0% CI is above 0%

3. Secondary Outcome: To Evaluate the Efficacy of HIL-214 Vaccine Against Moderate/Severe Acute Gastroenteritis (AGE) Associated With GI.1 or GII.4 Norovirus Genotypes, Irrespective of Other Gastrointestinal Pathogens.
Description: Time to first occurrence during the primary observation period* of moderate/severe AGE case associated with GI.1 or GII.4 norovirus genotypes, irrespective of other gastrointestinal pathogens. Vaccine efficacy (VE) is defined as 100% [1- (λV/λC)], where λV and λC denote the hazard rates of the primary endpoint AGE case for the HIL 214 and placebo arms, respectively. The primary endpoint AGE case is defined as at least 3 loose or liquid stools OR at least 2 or more episodes of vomiting OR 1 or more loose or liquid stools plus 1 or more vomiting episodes in any 24-hour period. The presence of norovirus in onset stool samples was assessed by RT-PCR and norovirus-positive samples were genotyped by sequencing.
Time Frame: The duration of the primary observation period was 6 months starting at 28 days post dose 2.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1399 | 1425
months | 3.11 (1.981) | 3.29 (1.628)
Statistical Analysis 1: Comparison: Placebo vs Experimental; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Vaccine Efficacy = 13.91, 95% CI 2-sided [-34.70 to 44.98] — Vaccine efficacy is demonstrated if the lower limit of the 95.0% CI is above 0%

4. Secondary Outcome: To Evaluate the Efficacy of HIL-214 Vaccine Against Moderate/Severe Acute Gastroenteritis (AGE) Associated With Any Norovirus Genogroup (GI or GII), Irrespective of Other Gastrointestinal Pathogens
Description: Time to first occurrence during the primary observation period of moderate/severe AGE case associated with any norovirus genogroup (GI or GII), irrespective of other gastrointestinal pathogens. Vaccine efficacy (VE) is defined as 100% [1- (λV/λC)], where λV and λC denote the hazard rates of the primary endpoint AGE case for the HIL 214 and placebo arms, respectively. The endpoint AGE case is defined as at least 3 loose or liquid stools OR at least 2 or more episodes of vomiting OR 1 or more loose or liquid stools plus 1 or more vomiting episodes in any 24-hour period. The presence of norovirus in onset stool samples was assessed by RT-PCR and norovirus positive samples were genogrouped by sequencing. Vaccine efficacy (VE) estimates and 95% confidence intervals (CIs) are also reported.
Time Frame: The duration of the primary observation period was 6 months starting at 28 days post dose 2.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1399 | 1425
months | 3.19 (1.852) | 3.17 (1.541)
Statistical Analysis 1: Comparison: Placebo vs Experimental; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Vaccine Efficacy = -6.37, 95% CI 2-sided [-45.04 to 22.00] — Vaccine efficacy is demonstrated if the lower limit of the 95.0% CI is above 0%

5. Secondary Outcome: Immunogenicity of HIL-214 Compared to Placebo
Description: The percentage of participants with a predefined seroresponse (≥4-fold rise in antibody concentration) at up to 56 days post dose 1 (Visit 2), 28 days post dose 2 (Visit 3), and/or at 1 year of age (visit 4) to the GI.1 and GII.4c components of HIL-214 and 95% confidence interval are reported. HBGA-blocking and pan-Ig assays were used for immunogenicity analyses
Time Frame: Participant reaches 1 year of age
Population: Full-Analysis Set, The FAS will include all subjects who are randomized and received at least 1 dose of HIL-214 or placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1538 | 1540
percentage of participants
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 2: number analyzed (Participants) | 1412 | 1445
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 2 | 0.6 [0.3 to 1.2] | 36.8 [34.3 to 39.4]
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 3: number analyzed (Participants) | 1390 | 1414
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 3 | 1.4 [0.8 to 2.1] | 95.5 [94.3 to 96.6]
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 4: number analyzed (Participants) | 1371 | 1391
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 4 | 1.6 [1.0 to 2.4] | 86.2 [84.3 to 88.0]
  Anti-GII.4c HBGA-blocking seroresponse rate at Visit 2: number analyzed (Participants) | 1412 | 1450
  Anti-GII.4c HBGA-blocking seroresponse rate at Visit 2 | 1.3 [0.8 to 2.1] | 7.4 [6.1 to 8.9]
  Anti- GII.4c HBGA-blocking seroresponse rate at Visit 3: number analyzed (Participants) | 1390 | 1416
  Anti- GII.4c HBGA-blocking seroresponse rate at Visit 3 | 2.2 [1.5 to 3.2] | 43.0 [40.4 to 45.6]
  Anti- GII.4c HBGA-blocking seroresponse rate at Visit 4: number analyzed (Participants) | 1371 | 1399
  Anti- GII.4c HBGA-blocking seroresponse rate at Visit 4 | 6.2 [5.0 to 7.6] | 25.0 [22.8 to 27.4]
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 2: number analyzed (Participants) | 1412 | 1450
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 2 | 0 [0.0 to 0.3] | 4.8 [3.7 to 6.0]
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 3: number analyzed (Participants) | 1390 | 1416
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 3 | 0.3 [0.1 to 0.7] | 42.3 [39.7 to 44.9]
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 4: number analyzed (Participants) | 1372 | 1400
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 4 | 0.2 [0.0 to 0.6] | 22.9 [20.7 to 25.2]
  Anti-GI.1 pan-Ig seroresponse rate at Visit 2: number analyzed (Participants) | 1411 | 1447
  Anti-GI.1 pan-Ig seroresponse rate at Visit 2 | 1.3 [0.8 to 2.1] | 84.6 [82.6 to 86.4]
  Anti-GI.1 pan-Ig seroresponse rate at Visit 3: number analyzed (Participants) | 1390 | 1414
  Anti-GI.1 pan-Ig seroresponse rate at Visit 3 | 2.4 [1.6 to 3.3] | 98.9 [98.3 to 99.4]
  Anti-GI.1 pan-Ig seroresponse rate at Visit 4: number analyzed (Participants) | 1371 | 1397
  Anti-GI.1 pan-Ig seroresponse rate at Visit 4 | 8.7 [7.2 to 10.3] | 97.1 [96.0 to 97.9]
  Anti-GII.4c pan-Ig seroresponse rate at Visit 2: number analyzed (Participants) | 1410 | 1448
  Anti-GII.4c pan-Ig seroresponse rate at Visit 2 | 3.3 [2.5 to 4.4] | 37.9 [35.4 to 40.5]
  Anti-GII.4c pan-Ig seroresponse rate at Visit 3: number analyzed (Participants) | 1390 | 1416
  Anti-GII.4c pan-Ig seroresponse rate at Visit 3 | 8.1 [6.7 to 9.7] | 83.9 [81.9 to 85.8]
  Anti-GII.4c pan-Ig seroresponse rate at Visit 4: number analyzed (Participants) | 1371 | 1398
  Anti-GII.4c pan-Ig seroresponse rate at Visit 4 | 23.6 [21.4 to 26.0] | 75.5 [73.1 to 77.7]
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate at Visit 2: number analyzed (Participants) | 1411 | 1448
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate at Visit 2 | 0.3 [0.1 to 0.7] | 35.9 [33.4 to 38.4]
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate at Visit 3: number analyzed (Participants) | 1390 | 1416
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate at Visit 3 | 1.0 [0.6 to 1.7] | 83.5 [81.4 to 85.4]
  Anti- GI.1 and GII.4c pan-Ig seroresponse rate at Visit 4: number analyzed (Participants) | 1371 | 1398
  Anti- GI.1 and GII.4c pan-Ig seroresponse rate at Visit 4 | 4.7 [3.7 to 6.0] | 74.7 [72.3 to 76.9]

6. Secondary Outcome: Safety of HIL-214 Compared to Placebo - Solicited Local Adverse Events (AEs)
Description: Percentage of participants with solicited local (injection site) adverse events (AEs) within 7 days of vaccine administration. Assessed AEs include injection site pain, erythema, induration, and swelling.
Time Frame: Up to 7 days after each dose of HIL-214 or placebo.
Population: Safety Analysis Set, all participants who were randomized and received at least 1 dose of trial vaccine (HIL-214 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1536 | 1541
percentage of participants
  Any solicited local AE | 6.7 | 10.4
  Injection site pain | 5.4 | 8.2
  Erythema | 1.8 | 2.0
  Induration | 0 | 0.7
  Swelling | 0.1 | 0.5

7. Secondary Outcome: Safety of HIL-214 Compared to Placebo - Solicited Systemic Adverse Events (AEs)
Description: Percentage of participants with solicited systemic AEs within 7 days of vaccine administration. Assessed AEs include drowsiness, irritability/fussiness, loss of appetite, vomiting, and diarrhea.
Time Frame: Up to 7 days after each dose of HIL-214 or placebo.
Population: Safety Analysis Set, all participants that received at least 1 dose of HIL-214 or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1536 | 1541
percentage of participants
  Any solicited systemic AE | 35.2 | 37.7
  Drowsiness | 10.7 | 12.7
  Irritability/fussiness | 18.0 | 20.2
  Loss of appetite | 7.9 | 8.4
  Vomiting | 7.4 | 8.6
  Diarrhea | 14.6 | 15.4

8. Secondary Outcome: Safety of HIL-214 Compared to Placebo - Adverse Events (AEs) Leading to Vaccine Withdrawal
Description: Percentage of participants with AEs leading to trial vaccine dose withdrawal.
Time Frame: Up to 28 days after first dose of HIL-214 or placebo.
Population: Safety Analysis Set; all participants that received at least 1 dose of HIL 214 or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1536 | 1541
percentage of participants | 0 | 0.1

9. Secondary Outcome: Safety of HIL-214 Compared to Placebo - Adverse Events (AEs) Leading to Trial Withdrawal.
Description: Percentage of participants with AEs leading to trial withdrawal.
Time Frame: From Day 1 to end of the trial/early termination.
Population: Safety Analysis Set; all participants that received at least 1 dose of HIL-214 or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 1536 | 1541
percentage of participants | 0.1 | 0.1

ADVERSE EVENTS:
Time Frame: Deaths from Day 1 to the end of 6 month observation period; Serious adverse events from Day 1 to the end of the trial; Unsolicited adverse events for up to 28 days after any dose of trial vaccine.
Description: Serious adverse events that occurred are reported at the preferred term level in the safety analysis set.
Arm/Group | Placebo | Experimental
All-Cause Mortality (participants affected / at risk) | 1/1536 | 2/1541
Serious Adverse Events (participants affected / at risk) | 165/1536 | 169/1541
Other Adverse Events (participants affected / at risk) | 889/1536 | 902/1541
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1536) | Experimental (N=1541)
Pneumonia (Infections and infestations) | 46 | 55
Bronchiolitis (Infections and infestations) | 23 | 35
Gastroenteritis (Infections and infestations) | 11 | 11
Pneumonia viral (Infections and infestations) | 5 | 5
Abscess limb (Infections and infestations) | 5 | 3
Amoebic dysentery (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 4 | 4
Burns second degree (Injury, poisoning and procedural complications) | 6 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Febrile convulsion (Nervous system disorders) | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 11 | 6
Anemia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 1
Sickle cell anemia (Congenital, familial and genetic disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 2
Pelvic mass (General disorders) | 1 | 0
Sudden infant death syndrome (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Dengue fever (Infections and infestations) | 4 | 5
Bronchitis (Infections and infestations) | 3 | 2
Atypical pneumonia (Infections and infestations) | 0 | 4
Cellulitis (Infections and infestations) | 2 | 2
Metapneumovirus bronchiolitis (Infections and infestations) | 1 | 2
Periorbital cellulitis (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 3 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 3
Chest wall abscess (Infections and infestations) | 1 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Adenovirus infection (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Giardiasis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Meningitis herpes (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Exposure via ingestion (Injury, poisoning and procedural complications) | 1 | 1
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 2
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Underweight (Metabolism and nutrition disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 2
Brain injury (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Intestinal anastomosis (Surgical and medical procedures) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Abscess of external ear (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0
Infection parasitic (Infections and infestations) | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Tethered oral tissue (Congenital, familial and genetic disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Post-procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1
Cholinergic syndrome (Nervous system disorders) | 0 | 1
Patient device incompatibility (Product Issues) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1536) | Experimental (N=1541)
Nasopharyngitis (Infections and infestations) | 474 | 492
Gastroenteritis (Infections and infestations) | 268 | 285
Upper respiratory tract infection (Infections and infestations) | 75 | 69
Bronchiolitis (Infections and infestations) | 39 | 47
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 55 | 64
Diarrhea (Gastrointestinal disorders) | 40 | 31
Anemia (Blood and lymphatic system disorders) | 30 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT05281094/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT05281094/SAP_001.pdf